CLINICAL TRIAL: NCT02957981
Title: The Genetic Education for Men (GEM) Trial: Web-Based Genetic Education vs. Standard Care in Men From Hereditary Cancer Families
Brief Title: The Genetic Education for Men Trial: Web-Based Education vs. Standard Care
Acronym: GEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Marc D Schwartz, Professor of Oncology, Associate Director for Population Science, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-1162
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Prostate Carcinoma; Breast Neoplasm; Pancreatic Cancer; BRCA1 Mutation; BRCA2 Mutation
Keywords: BRCA1; BRCA2; Men; Hereditary Cancer; Prostate Cancer; Male Breast Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Multiple Endocrine Neoplasia Type 1; Breast Neoplasms, Male | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Counseling (Experimental): Genetic information provided via an individually tailored website.
  Interventions: Behavioral: Web-based Counseling
- Standard Care (Active Comparator): Participants are not provided with web-based education but can choose to pursue genetic counseling and testing.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Web-based Counseling — The web-based genetic counseling and education intervention will include standard information typically provided in individual genetic counseling. the intervention will be individually tailored based upon key clinical and demographic characteristics of the participant.
  Arms: Web-Based Counseling
Behavioral: Standard Care — Standard care includes access to resource list for men from hereditary cancer families plus access to standard clinical genetic counseling
  Arms: Standard Care

SUMMARY:
The primary goal of this research is to develop and test a web-based genetic education/counseling intervention. This intervention is designed to educate men from hereditary cancer families about the personal relevance of genetic testing in order to help them make decisions about whether to pursue genetic testing. The investigators will test this intervention against standard care for men from hereditary cancer families. The web-based educational intervention includes all of the information typically covered during genetic counseling. As a result, after completing the education intervention participants can proceed directly to genetic testing if they choose. The investigators will conduct a survey prior to randomization and then follow-up surveys at 1-month and 6-months post-randomization. The primary outcome will be uptake of genetic testing. Secondary outcomes will be completion of genetic counseling and decision satisfaction.

DETAILED DESCRIPTION:
Aim 1: Develop a web-based intervention to increase genetic counseling/testing uptake in men at high risk for carrying a BRCA mutation.

Aim 2: Evaluate the impact of the web-based intervention (WI) vs. usual care (UC)

Aim 3: Examine the behavioral and psychosocial impact of BRCA testing in men from BRCA families.

Identification and Recruitment of Subjects. Participants will be recruited via the Lombardi Comprehensive Cancer Center's Familial Cancer Registry and the Non-therapeutic Subject Registry Shared Resource. These registries contain over 800 female BRCA1/2 positive participants. In addition, the investigators will recontact participants from prior trials who have consented to be recontacted for future research and will accept self-referred index cases who contact the study about participation. Female index cases will be identified based on vital status, recency of contact, and availability of test reports documenting their positive BRCA1/2 status. Where available, pedigrees will also be reviewed.

To protect the privacy of study participants, participants will be recruited through their female BRCA mutation carrier relatives (index patients) who will provide their contact information. The investigators will identify adult female mutation carriers who are enrolled in the Non-therapeutic Subject Registry Shared Resource, Familial Cancer Registry, who received a positive test result as a participant in IRB 2004-133 and provided consent to be contacted about future research studies or who contact the study directly about enrollment. The study staff will mail a study invitation to potentially eligible index cases. This mailing will include: an introductory letter; an informed consent document; a HIPAA Authorization form; study brochures for distribution to male relatives if desired; and a family contact form requesting contact information and current ages for potentially eligible male relatives. The investigators will request that index patients return the Family Contact Form in a self-addressed stamped envelope or complete an electronic version of the form. Consistent with prior research and Institutional Review Board guidance, the letter and Family Contact Form will reiterate that index patients should request permission from their potentially eligible male relative(s) prior to providing contact information to us, and the index patient's signature on the Family Contact Form will attest to this. The packet will also contain information on how women may decline participation (an opt-out post card). If, after 2-3 weeks, individuals do not decline participation, a research assistant will call to determine interest in the study and request completion of the Family Contact Form.

Upon receiving returned Family Contact Forms, the research team we will contact potentially eligible male relatives by mail. The study packet that is sent will include: an introductory letter; informed consent document; study brochure, and opt-out postcard. On the opt-out contacts, men can also indicate if they are ineligible for the study due to a cancer diagnosis or prior genetic counseling/testing.

Baseline survey. The baseline survey can be completed via telephone or electronically. Two weeks following the mailing, the researchers will contact eligible men who have not opted out by email or telephone. For email contact, the investigators will send an email link to an electronic study consent and baseline survey. If no email address is provided, a research assistant will contact the participant by telephone. If the participant has already returned the print informed consent document, the research assistant will answer any questions about the study and proceed with the baseline survey. If the participant has not returned an informed consent document, the research assistant will complete a verbal consent process and administer the baseline survey.

Randomization. Following completion of the baseline survey, a research assistant will randomize participants to either the Web Intervention or Usual Care. Randomization will be achieved via computer generated random numbers (blocks of 8). Family members will be assigned to the same intervention to avoid contamination. Men who complete the baseline survey online will be notified of their randomization assignment via email. Men who complete the baseline survey by telephone will be notified of their randomization status at the end of the baseline survey.

Usual Care Group. Men who are randomized to the Usual Care arm will receive an email and letter informing them of their group assignment. These contacts will include a list of resources for men from hereditary cancer families and for those who have not previously completed the print or electronic consent form, another copy of the print consent and a link to the electronic consent will also be provided. At this time, Usual Care participants will be informed that if they are interested in genetic counseling and testing, they can contact the study team (via a toll-free number provided to them in the letter) to schedule a telephone genetic counseling session (free of charge) or the study team can provide a local referral for in-person genetic counseling. All participants will be required to complete the print or electronic study consent form prior to study-provided genetic counseling.

Web Intervention Group. Men randomized to the Web Intervention will receive an email and letter (sent through US Mail) with the web address, and an individualized code. When participants access the website, they will be asked to enter their email address and their code, and then choose a password for future log-ins. Participants who forget their passwords can request a new log-in code at any time. The investigators will provide participants with a toll-free support number to call if they have any questions. Participants who have not completed the print or electronic informed consent document will be required to complete the electronic consent prior to viewing the Web Intervention.

At the conclusion of the Web Intervention, participants will be provided with the following options for pursuing genetic testing for their familial BRCA1 or BRCA2 mutation: 1) they can indicate that they are not interested in pursuing genetic testing; 2) they can indicate that they have questions about genetic testing, in which case an RA will follow-up, answer any process-related questions, and determine if a genetic counselor consultation is required; 3) they can schedule an individual genetic counseling session (with a LCCC genetic counselor or with a genetic counselor of their choice); 4) they can proceed directly to genetic testing.

Pre-Test Genetic counseling. All participants have multiple options for pre-test genetic counseling. Since the Web Intervention provides participants with content that is comparable to that of standard pre-test genetic counseling, Web Intervention participants have the option to proceed directly to genetic testing after viewing the intervention. However, since we expect that some participants may prefer traditional genetic counseling, participants will have the option of free pre-test telephone genetic counseling provided through the study by a board-certified genetic counselor at the Lombardi Comprehensive Cancer Center. In contrast, because Usual Care participants will not receive electronic genetic education/counseling, they will not have the option to proceed directly to genetic testing. Usual Care participants who are interested in pursuing genetic counseling will have the option to receive free pre-test telephone genetic counseling through the study by a board certified genetic counselor at Lombardi Comprehensive Cancer Center. After completing genetic counseling, participants will be provided with the opportunity to proceed to genetic testing. This arm is designed to replicate standard care in which individual genetic counseling often proceeds genetic testing.

Men in either group who prefer in-person genetic counseling, will be provided with a referral to a local counselor and informed that those costs are not covered by the study. Men whose insurance company requires them to be seen by a genetic counselor within a specified organization before testing is ordered will be informed of that requirement if they proceed to testing.

Genetic testing. Genetic testing is not required as part of this study. Any participants interested in proceeding with genetic testing will receive standard clinical genetic testing from a certified commercial laboratory. All testing will be provided under standard clinical protocols and laboratory consents. The standard of care for relatives of BRCA1 or BRCA2 carriers is to test only for the specific familial mutation. The familial mutation will be known to study staff because documentation of test reports must be available for female cases, from whom eligible participants for the study are recruited. Men who have Ashkenazi Jewish background will be offered testing for the three BRCA mutations common in this ethnic group, as is also standard clinical practice. Men will have the option to go through their insurance company or pay out of pocket for genetic testing. In either case, the fees associated with testing will be paid directly to the clinical laboratory that performs the test.

Coordination of genetic testing. All participants who indicate that they are interested in genetic testing will be contacted by a research assistant to obtain information needed for insurance billing, pre-verification and the completion of laboratory test requisition forms. The research assistant will provide a laboratory consent form and laboratory requisition form to participants who are interested in completing genetic testing. After these completed and signed forms are returned to us, the research assistant will send the participant a kit to collect saliva (DNA). The participant is then responsible for mailing the postage paid DNA kit and required forms directly to the testing laboratory. Billing and payment arrangements for testing will be handled between the testing lab and the participant. Georgetown University will not bill patients for genetic testing services.

Post-test genetic counseling. All participants who receive genetic testing through the study will receive individual post-test genetic counseling by telephone from a board-certified genetic counselor. In general, DNA testing results are available within 2 weeks. Results will be sent directly to a study genetic counselor. The genetic counselor will call the participant to review the test results, including cancer risks, management options/guidelines, implications to family members, and emotional response to testing. Questions and concerns will be addressed, and referrals for follow-up will be provided as needed, including (if appropriate), genetic counseling referrals for relatives. If participants did not undergo pre-test genetic counseling, a brief medical and family history will be taken at this time, so that risk and management information can be individualized. This session is expected to take between 10 to 30 minutes.

After the post-test session, the genetic counselor will mail a copy of the laboratory's genetic testing report and a brief genetic counseling summary letter that the participant can share with his health care providers and family members if desired.

Follow-Up Survey. Participants will be contacted for follow-up surveys at 1-month and 6-months post-randomization. These surveys will be similar to (but shorter than) the baseline survey. As for the baseline survey, these follow-up surveys will be conducted electronically or via telephone. Participants who have provided verbal consent at the time of the baseline but who have not completed written or electronic consent (and therefore have not proceeded to genetic counseling) will remain eligible to complete the follow-up surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age 25 -70
3. At least one first-, or second--degree relative who has been found to carry a BRCA1 or BRCA2 mutation.

Exclusion Criteria:

1. Personal diagnosis of any cancer, other than non-melanoma skin cancer
2. Prior genetic counseling or testing for hereditary breast/ovarian cancer
3. Family history suggestive of a hereditary cancer syndrome not attributable to the BRCA1 or BRCA2 mutation in their family, based on pedigree review by the study team
4. An uncertain risk of carrying the familial BRCA1 or BRCA2 mutation (e.g., because it is not clear on what side of the family the mutation is segregating), based on pedigree review by the study team
5. Have one one or more children who are BRCA1 or BRCA2 positive
6. Cannot participate in or understand English
7. Cannot provide meaningful informed consent

Ages: 25 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Completion of BRCA1/BRCA2 Gene Testing | 6-months
  The number of participants in each arm who choose to be tested for the BRCA1 or BRCA2 mutation that has previously been identified in their family.

SECONDARY OUTCOMES:
Completion of Genetic Counseling | 6-months
  The number of men in each arm who choose to obtain genetic counseling
Decision Satisfaction | 6-Months
  Scores on the satisfaction with decision scale at 6-months post-randomization
Decision Conflict | 6-Months
  Scores on the decision conflict scale at 6-months post-randomization

OTHER OUTCOMES:
Cancer Distress | 6-Months
  Impact of Events Scale
Genetic Testing Distress | 6-Months
  Multidimensional Impact of Cancer Risk Assessment Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center/Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared with other researchers.

REFERENCES:
- [Derived] Grisham C, Peshkin BN, Sorgen L, Isaacs C, Ladd MK, Jacobs A, Binion S, Tynan M, Kuchinsky E, Friedman S, Taylor KL, Graves K, O'Neill S, Kim D, Schwartz MD. Streamlined Genetic Education and Cascade Testing in Men from Hereditary Breast Ovarian Cancer Families: A Randomized Trial. Public Health Genomics. 2024;27(1):100-109. doi: 10.1159/000540466. Epub 2024 Aug 22. PMID 39173603